CLINICAL TRIAL: NCT00727597
Title: A Study in Underrepresented Patient Population or Regimen Tolerability: SUPPoRT
Acronym: SUPPoRT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Princy Kumar, MD, Principal Investigator, Georgetown University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL 110408
Record Dates: First submitted 2008-07-31; First posted 2008-08-04 (Estimated); Results first posted 2013-07-02 (Estimated); Last update posted 2013-07-02 (Estimated); Status verified 2013-06

CONDITIONS: Human Immunodeficiency Virus Infections
MeSH Terms: interventions — efavirenz; fosamprenavir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A : Boosted Lexiva plus Epzicom (Experimental): Once daily (QD) regimen of Lexiva (fosamprenavir 1400 mg) + Norvir (ritonavir 100 mg) + Epzicom (abacavir 600 mg / lamivudine 300 mg).
  Interventions: Drug: Boosted Lexiva
- Arm B: Efavirenz plus Epzicom (Experimental): QD regimen of Sustiva (efavirenz 600 mg) + Epzicom (abacavir 600 mg / lamivudine 300 mg)
  Interventions: Drug: Efavirenz 600mg

INTERVENTIONS:
Drug: Efavirenz 600mg — QD regimen of Sustiva (efavirenz 600 mg) + Epzicom (abacavir 600 mg / lamivudine 300 mg)
  The intervention may be switched for the following reasons:
  * To resolve a Grade 3 or 4 Adverse Event
  * The subject experienced a virologic failure (as defined in section 3.6.2)
  * The investigator believes the subject is at a significant risk for failing to comply with the protocol AND the investigator believes a regimen substitution is likely to resolve the compliance issue
  * The investigator believes there is any other significant safety concern for the subject associated with remaining on the current regimen (e.g., hypersensitivity reaction, increased risk of suicide)
  Other Names: Efavirenz(Sustiva)600 mg
  Arms: Arm B: Efavirenz plus Epzicom
Drug: Boosted Lexiva — Once daily (QD) regimen of Lexiva (fosamprenavir 1400 mg) + Norvir (ritonavir 100 mg) + Epzicom (abacavir 600 mg / lamivudine 300 mg)
  The intervention may be switched for the following reasons:
  * To resolve a Grade 3 or 4 Adverse Event
  * The subject experienced a virologic failure (as defined in section 3.6.2)
  * The investigator believes the subject is at a significant risk for failing to comply with the protocol AND the investigator believes a regimen substitution is likely to resolve the compliance issue
  * The investigator believes there is any other significant safety concern for the subject associated with remaining on the current regimen (e.g., hypersensitivity reaction, increased risk of suicide)
  Other Names: Fosamprenavir(Lexiva)
  Arms: Arm A : Boosted Lexiva plus Epzicom

SUMMARY:
The hope of this study is to gather data and information about the tolerability and effectiveness of Lexiva versus Sustiva in patients who have have been generally underrepresented in clinical trials.

DETAILED DESCRIPTION:
The objective of this study is to gain tolerability and efficacy data for Norvir-boosted Lexiva versus Sustiva, both used in combination with Epzicom, as components of a first-line, once daily regimen for the treatment of HIV-1 infection in a patient population that is underrepresented in US clinical research.

ELIGIBILITY:
Inclusion Criteria:

Screening plasma HIV-1 RNA viral load >5000 copies/mL Self-identification as having any non-White/Caucasian European geographic ancestry (i.e., an individual is eligible if she/he does not have any White/Caucasian European ancestry; OR an individual is eligible if she/he indicates a mix of White/Caucasian European ancestry AND one or more other geographic ancestries); Antiretroviral-naïve (no treatment with any antiretroviral drug in the 28 days prior to study entry and ≤14 days of treatment ever with any antiretroviral drug) Negative test for the HLA-B*5701 allele Ability and willingness to give written informed consent

Either gender is eligible, but enrollment of at least two female subjects to every one male subject is strongly encouraged. A female subject is eligible to participate in the study if she is of:

1. Non-childbearing potential or,
2. Childbearing potential with a negative pregnancy test at screen and agrees to use one of the following methods of contraception:

i. Agreement for complete abstinence from intercourse from 2 weeks prior to administration of investigational products, throughout the study, and for 2 weeks after discontinuation of all study medications; ii. Double barrier contraception (male condom/spermicide, male condom/diaphragm, diaphragm/spermicide); iii. Any intrauterine device (IUD) with published data showing that the expected failure rate is less than 1% per year (not all IUDs meet this criterion); iv. Any other method with published data showing that the lowest expected failure rate for the method is less than 1% per year. v. Sterilization (female subject or male partner of female subject)

Exclusion Criteria:

Screening HIV-1 genotype indicating the presence of any of the following mutations in the reverse transcriptase (RT) region: K65R, L74V, K103N, Y115F, Y181C/I, Y188C/L/H or G190S/A, or a combination of two or more thymidine analog mutations (M41L, D67N, K70R, K219Q or E) that include changes at either L210 or T215, associated with resistance to abacavir, lamivudine, or efavirenz; OR within the protease region, detection of any of the following mutations associated with resistance to fosamprenavir or ritonavir: I50V, I54L/M, I84V, or the combination of the two mutations V32I+I147V Positive for Hepatitis B surface antigen (HBsAg+)

Requirement for active treatment for hepatitis C virus infection, as indicated by both a positive Hepatitis C Virus serology AND either:

1. Decompensated liver disease, or
2. Aspartate aminotransferase (AST) >3X the upper limit of normal (ULN), or
3. Alanine aminotransferase (ALT) >3X the ULN Currently pregnant, intending to become pregnant during the study period, or breast-feeding Use of immunomodulators (e.g., interleukins, interferons, cyclosporine), any vaccinations, systemic cytotoxic chemotherapy, or investigational therapy within 28 days prior to study entry. Chronic treatment with prednisone at a daily dose of 10 mg or less is permitted. Acute treatment (less than 21 days) with larger doses of corticosteroids for acute therapy is permitted.

Active or suspected drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements Judged by the investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results Active or acute Centers for Disease Control Clinical Category C event at screening. (Note: Treatment for the acute event must have been completed at least 28 days prior to screening.) Clinically relevant pancreatitis or clinically relevant hepatitis at screening Hgb<8g/dl, platelet count <50,000/mm3, calculated creatinine clearance <50ml/min via Cockroft-Gault equation, or AST or ALT > 5X the ULN Any Grade 4 laboratory abnormality

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2008-07; Primary Completion 2010-08 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Princy Kumar, MD, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University, Washington D.C., District of Columbia, United States

REFERENCES:
- [Derived] Kumar P, DeJesus E, Huhn G, Sloan L, Small CB, Edelstein H, Felizarta F, Hao R, Ross L, Stancil B, Pappa K, Ha B; SUPPORT Study Team. Evaluation of cardiovascular biomarkers in a randomized trial of fosamprenavir/ritonavir vs. efavirenz with abacavir/lamivudine in underrepresented, antiretroviral-naive, HIV-infected patients (SUPPORT): 96-week results. BMC Infect Dis. 2013 Jun 7;13:269. doi: 10.1186/1471-2334-13-269. PMID 23741991

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients ≥18 years of age who were ART-naïve (≤14 days of treatment with any ART agent), HLA-B*5701-negative, and had a screening HIV-1 RNA >5000 copies/mL. Patients were required to be of minority race or ethnicity; white, non-Hispanic patients were not eligible for this study.
Groups:
- Once Daily (QD) Regimen of Lexiva: Once daily (QD) regimen of Lexiva (fosamprenavir 1400 mg) + Norvir (ritonavir 100 mg) + Epzicom (abacavir 600 mg / lamivudine 300 mg).
- QD Regimen of Sustiva: QD regimen of Sustiva (efavirenz 600 mg) + Epzicom (abacavir 600 mg / lamivudine 300 mg)
Period: Overall Study
Arm/Group | Once Daily (QD) Regimen of Lexiva | QD Regimen of Sustiva
Started | 51 | 50
Completed | 51 | 50
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Once Daily (QD) Regimen of Lexiva | QD Regimen of Sustiva | Total
Number analyzed (Participants) | 51 | 50 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 1 | 0 | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 33.5 (2) | 34 (2) | 34 (2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 35 | 34 | 69
Region of Enrollment [Number; unit: participants]
  United States | 51 | 50 | 101

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Needing to Switch Comparator Drugs (FPV/r or EFV)
Description: Subjects were randomized and initiated treatment on one of the antiretroviral arms(FPV/r or EFV) at study Entry visit. Subjects would be switched for the follwing reasons:
  * To resolve a Grade 3 or 4 Adverse Event
  * The subject experienced a virologic failure (as defined in section 3.6.2)
  * The investigator believes the subject is at a significant risk for failing to comply with the protocol AND the investigator believes a regimen substitution is likely to resolve the compliance issue
  * The investigator believes there is any other significant safety concern for the subject associated with remaining on the current regimen (e.g., hypersensitivity reaction, increased risk of suicide)
Time Frame: 96 weeks
Measure: Number; unit: participants
Arm/Group | Once Daily (QD) Regimen of Lexiva | QD Regimen of Sustiva
Number analyzed (Participants) | 51 | 50
participants | 1 | 2

2. Primary Outcome: Number of Subjects Developing Any Treatment-related Grade 3-4 Adverse Events
Time Frame: 96 weeks
Measure: Number; unit: participants
Arm/Group | Once Daily (QD) Regimen of Lexiva | QD Regimen of Sustiva
Number analyzed (Participants) | 51 | 50
participants | 2 | 3

ADVERSE EVENTS:
Arm/Group | Once Daily (QD) Regimen of Lexiva | QD Regimen of Sustiva
Serious Adverse Events (participants affected / at risk) | 2/51 | 2/50
Other Adverse Events (participants affected / at risk) | 9/51 | 15/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once Daily (QD) Regimen of Lexiva (N=51) | QD Regimen of Sustiva (N=50)
Cardiac Arrest (Cardiac disorders) | 1 (1) | 0 (0)
Suspected Drug Hypersensitivity to ABC (Immune system disorders) | 1 (1) | 1 (1)
Acute Pancreatitis (Endocrine disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Once Daily (QD) Regimen of Lexiva (N=51) | QD Regimen of Sustiva (N=50)
cholesterol, total neutrophils, creatine kinase, and triglycerides (General disorders) | 9 (9) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No